CLINICAL TRIAL: NCT01214577
Title: A Phase 2a, Multi-Centre, Single Arm Study to Evaluate the Safety and Efficacy of PEP005(Ingenol Mebutate) Gel, 0.015%, in Patients With Photo-damaged Skin on the Face
Brief Title: Study to Evaluate the Safety and Efficacy of PEP005 (Ingenol Mebutate) Gel, 0.015%, in Patients With Photo-damaged Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Jacqueline Morley, Clinical Research Team Leader, Peplin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-036
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Photo-damage
Keywords: PEP005; Peplin; Photo-damage
MeSH Terms: interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Up to three days of treatment
  Interventions: Drug: PEP005 (ingenol mebutate) Gel

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel — 0.015%

SUMMARY:
This study is primarily designed to evaluate the safety and tolerability of PEP005 Gel, 0.015% when administered for up to three consecutive days to photo-damaged skin on the face. The secondary endpoint is to determine the efficacy of PEP005 Gel, 0.015% when administered for up to three consecutive days in patients with photo-damaged skin on the face.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients aged 30 to 65 years.
2. Female patients must be of either:

   * Non-childbearing potential, provided there is a laboratory confirmed serum follicle stimulating hormone (FSH) level ≥ 40mIU/ml or there is a confirmed clinical history of sterility (e.g., the patient is without a uterus); or
   * Childbearing potential, provided there are negative urine pregnancy test results prior to study treatment, to rule out pregnancy.
3. Patient has provided informed consent documented by signing the Informed Consent Form (ICF) prior to any study-related procedures, including any alteration of medications in preparation for study entry.
4. Patient has agreed to allow photographs of the selected treatment area to be taken and used as part of the study data package.

Exclusion Criteria

1. Known sensitivity or allergy to any of the ingredients in PEP005 (ingenol mebutate) Gel.
2. Current enrolment or participation in a clinical research study within 30 days of entry into this study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of PEP005 Gel, 0.015% when administered for up to three consecutive days to photo-damaged skin on the face. | Day 43

SECONDARY OUTCOMES:
To determine the efficacy of PEP005 Gel, 0.015% when administered for up to three consecutive days in patients with photo-damaged skin on the face. | Day 43

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - The Skin Centre, Benowa, Queensland
  - Specialist Connect, Woolloongabba, Queensland

REFERENCES:
- See also: Related Info — http://www.tga.gov.au/